CLINICAL TRIAL: NCT04576663
Title: Phenylephrine Prophylaxis for Postspinal Anesthesia Hypotension in Parturients With Preeclampsia Undergoing Cesarean Section: a Randomized, Placebo-controlled Dose-finding Trial
Brief Title: Phenylephrine Prophylaxis for Postspinal Anesthesia Hypotension in Parturients With Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Yi Chen-2020-6
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-09

CONDITIONS: Adverse Effect
Keywords: Phenylephrine; Postspinal anesthesia hypotension; Preeclampsia; Cesarean section; Dose-finding
MeSH Terms: conditions — Pre-Eclampsia | interventions — Saline Solution; Phenylephrine; Vasoconstrictor Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Placebo Comparator): Normal saline infusion simultaneous with subarachnoid block
  Interventions: Drug: Normal saline
- 0.3125 μg/kg/min group (Experimental): A maintenance dose of phenylephrine (0.3125 μg/kg/ min) infusion simultaneous with subarachnoid block
  Interventions: Drug: Phenylephrine
- 0.625 μg/kg/min group (Experimental): A maintenance dose of phenylephrine (0.625 μg/kg/ min) infusion simultaneous with subarachnoid block
  Interventions: Drug: Phenylephrine
- 0.9375 μg/kg/min group (Experimental): A maintenance dose of phenylephrine (0.9375 μg/kg/ min) infusion simultaneous with subarachnoid block
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Normal saline — Normal saline infusion simultaneous with subarachnoid block
  Other Names: NS
  Arms: Control group
Drug: Phenylephrine — Different infusion dose of phenylephrine simultaneous with subarachnoid block
  Other Names: Vasopressors
  Arms: 0.3125 μg/kg/min group; 0.625 μg/kg/min group; 0.9375 μg/kg/min group

SUMMARY:
The purpose of this study is to investigate the suitable infusion dose of phenylephrine for prophylaxis against postspinal anesthesia hypotension in parturients with preeclampsia undergoing cesarean section.

DETAILED DESCRIPTION:
Preeclampsia, which affects 5% to 7% of parturients, is a significant cause of maternal and neonatal morbidity and mortality. Because of constricted myometrial spiral arteries with exaggerated vasomotor responsiveness, though blood pressure in parturients with preeclampsia are apparently higher than healthy parturients, placental hypoperfusion is more common. Spinal anesthesia is still the preferred mode of anesthesia in parturients with preeclampsia for cesarean section. In preeclampsia parturients, spinal anesthesia improve intervillous blood flow (provided that hypotension is avoided) which contribute to increase placental perfusion. Even so, 17-26% parturients with preeclampsia experienced postspinal anesthesia hypotension due to the extensive sympathetic block that occurred with spinal anesthesia. Practical guidelines for obstetric anesthesia from the American Society of Anesthesiologists and an international consensus statement on the management of hypotension with vasopressors indicate either IV ephedrine or phenylephrine may be used to correct hypotension. But the suitable infusion dose of phenylephrine in parturients with preeclampsia is still unknown. The purpose of this study is to investigate the suitable infusion dose of phenylephrine for prophylaxis against post-spinal anesthesia hypotension in parturients with preeclampsia undergoing cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥32 weeks
* American Society of Anesthesiologists physical status classification II to III
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Baseline blood pressure ≥180 mmHg
* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-09-21 (Estimated)

PRIMARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 80% of the baseline

SECONDARY OUTCOMES:
Overall stability of systolic blood pressure control versus baseline | 1-15 minutes after spinal anesthesia
  Evaluated by performance error (PE)
Overall stability of heart rate control versus baseline | 1-15 minutes after spinal anesthesia
  Evaluated by performance error (PE)
The incidence of severe post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of nausea and vomiting | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of bradycardia | 1-15 minutes after spinal anesthesia
  Heart rate < 60 beats/min
The incidence of hypertension. | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery
  From umbilical arterial blood gases.
Partial pressure of oxygen | Immediately after delivery
  From umbilical arterial blood gases.
Base excess | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration
APGAR score | 5 min after delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration

CONTACTS AND LOCATIONS:
Overall Officials: Xinli Ni, Dr., Study Chair — Hospital of Ningxia Medical University